CLINICAL TRIAL: NCT05306977
Title: Open-label Pilot to Test a Novel 1 Hz Intensive Repetitive Transcranial Magnetic Stimulation Paradigm in Patients With Anxiety
Brief Title: rTMS Pilot for Anxiety
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: pilot project. grant not funded
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 850766
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Results first posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Intervention Model Description: Aim 1: Outcome measures. Anxiety potentiated startle (APS) Statistical Analysis. The main analysis will be a paired-sample t-test (pre vs. post stimulation).
  Aim 2: Outcome measures. Accuracy and reaction time during the visual short term memory task (VSTM). Statistical Analysis. The main analysis will be a 2 [stimulation: pre-stimulation vs. post-stimulation] by 2 [load: low vs. high] repeated-measures ANOVA. Safety and Adverse Events
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Pilot arm (Other): Aims 1 and 2 of this project will be tested using a within-subjects design where anxiety patients will receive a 5-day course of accelerated 1 Hz rTMS (8x session x 600 pulses/session) to the right IPS.
  Interventions: Device: Open-label accelerated 1 Hz repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Open-label accelerated 1 Hz repetitive transcranial magnetic stimulation — Patients will receive a 5-day course of accelerated 1 Hz rTMS (8x session x 600 pulses/session) to the right intraparietal sulcus. Subjects will receive a continuous train of 1 Hz stimulation. They will receive a total of 600 pulses per train. Trains will be separated by ~50 min rest intervals.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of 1 Hz parietal stimulation in anxiety. Our approach will be to administer 1 week of open-label accelerated 1 Hz parietal rTMS (5 days, 8 sessions/day, 600 pulses/session) and measure the effect of this neuromodulation on APS, and short term memory in a cohort of anxiety GAD patients.

DETAILED DESCRIPTION:
Aims 1 and 2 of this project will be tested using a within-subjects design where anxiety patients will receive a 5-day course of accelerated 1 Hz rTMS (8x session x 600 pulses/session) to the right IPS. In Aim 1, we will test the effects of this stimulation on arousal during the NPU threat task (NPU section). In Aim 2 below, we will test the effects of this stimulation on arousal-related attention control deficits using the VSTM task (VSTM section).

Subjects will undergo 7 study visits spaced over a roughly 3-week period depending upon availability. First, subjects will have a pre-stimulation test visit. On this visit they will undergo the following procedures: 1) motor threshold testing, 2) noise habituation, 3) shock workup 4) NPU task, 5) VSTM task. Then they will have 5 rTMS visits. On these visits, subjects will receive 8 trains of 1 Hz rTMS (600 pulses per train, each separated by ~50 min). Finally, they will have a post-stimulation test visit, which will included the noise habituation, shock workup, NPU task, and VSTM task.

ELIGIBILITY:
Inclusion Criteria

* Meet the DSM-V criteria for an anxiety disorder (i.e. generalized anxiety disorder, social anxiety disorder, panic disorder, etc.)
* Subjects must be 18-50 years old
* Able to give their consent
* Right-handed

Exclusion Criteria

* Non-english speaking
* Any significant medical or neurological problems
* Current or past (non-anxiety) Axis I psychiatric disorder(s), active or history of active suicidal ideation
* Alcohol/drug problems in the past year or lifetime alcohol or drug dependence
* Any medical condition that increases risk for TMS
* History of seizure
* History of epilepsy
* Increased risk of seizure for any reason
* Pregnancy, or positive pregnancy test
* Hearing loss

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas L Balderston, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

REFERENCES:
- [Background] Balderston NL, Beydler EM, Goodwin M, Deng ZD, Radman T, Luber B, Lisanby SH, Ernst M, Grillon C. Low-frequency parietal repetitive transcranial magnetic stimulation reduces fear and anxiety. Transl Psychiatry. 2020 Feb 17;10(1):68. doi: 10.1038/s41398-020-0751-8. PMID 32066739
- See also: Online Screening Form — https://is.gd/cndslab

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pilot Arm
Started | 5
Completed | 4
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pilot Arm
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.4 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Anxiety Potentiated Startle (APS)
Description: Electromyography (EMG) startle responses were recorded from the left orbicularis oculi muscle using a Biopac MP160 unit (Biopac; Goleta, CA) via 15 × 20 mm electrodes (Rhythmlink #DECUS10026; Columbia, SC).
  EMG was bandpass filtered from 30 to 300 Hz, rectified, and smoothed using a 20-ms sliding window. Startle responses were scored as the peak (max during the 20 ms to 120 ms post-noise window) - the baseline (50 ms pre-noise window), and converted to t-scores with a mean of 50 and a standard deviation of 10 (tx = [Zx × 10] + 50). Greater t-scores mean larger blinks, which could be associated with greater anxiety, however there is no clinically relevent threshold. Noisy trials (baseline SD > 2x run SD) were excluded, and "no blink" (peak < baseline range) trials were coded as 0. To calculate APS within each timepoint, we subtracted the response during the neutral ITI from the response during the unpredictable ITI. T-scores represent the change from baseline to post stimulation.
Time Frame: Post stimulation
Population: Outcome measures. Anxiety potentiated startle (APS) contrasted between pre and post stimulation
Measure: Mean (Standard Deviation); unit: T-score (pre - post)
Arm/Group | Pilot Arm
Number analyzed (Participants) | 4
T-score (pre - post) | 1.89 (3.54)

2. Primary Outcome: Visual Short Term Memory Performance (VSTM)
Description: Visual short term memory task: This task has been adapted from Vogel & Machizawa (Vogel & Machizawa, 2004). On each trial, subjects see an arrow (cue) pointing to the left or the right. After a short delay, they see a bilateral array of squares that vary in color, location, and angle of rotation (memory array). Subjects are instructed to encode the squares in the cued hemifield (targets) and ignore the squares contralateral to the cued hemifield (distractors). After another short delay (retention interval), subjects see a single square (response prompt) that is either an exact match (same color/location/angle) or a complete mismatch (different color/location/angle). Subjects are instructed to indicate whether the square is a match or a mismatch.
Time Frame: Pre and post stimulation
Population: Aim 2: Outcome measures. Reaction time during the visual short term memory task (VSTM) contrasted pre and pot stimulation.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Pilot Arm
Number analyzed (Participants) | 4
msec | -58.6 (495.1)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Pilot Arm
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT05306977/Prot_SAP_000.pdf